CLINICAL TRIAL: NCT01643317
Title: Screening Cardiovascular Patients for Aortic Aneurysms
Acronym: SCAN
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Joep Teijink, MD, PhD, Vascular Surgeon, Catharina Ziekenhuis Eindhoven
Other Study IDs: Catharina_Project_SCAN
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Screening studies for Abdominal Aortic Aneurysms (AAA) in 65 to 79 years aged men, have shown a significant reduction in AAA related mortality. In addition, the cost-effectiveness of screening for AAA in men in the Netherlands has been demonstrated by using a Markov model. Screening might be even more (cost-) effective if targeted on high risk groups, such as patients with a particular cardiovascular disease with a known increased risk of having an AAA.

Project SCAN (Screening CardioVascular patients for Aortic aNeurysms) is a project focused on targeted AAA screening to proactively diagnose patients at high risk of having an aneurysm that eventually may rupture. This pilot project aims to study the value of a screening protocol in daily practice to detect AAA's in high risk patients.

DETAILED DESCRIPTION:
1. Offering PAD and CAD patients a non-invasive abdominal ultrasound after a careful process of shared-decision making
2. Recording data on aneurysm detection on all PAD and CAD patients screened:

   1. General information (age, gender)
   2. Medical history on CardioVascular risk factors (such as smoking history, hypertension, and other cardiovascular medical conditions - only information that is already recorded in the patient's medical history chart)
   3. AAA - Yes/ No (Yes if ≥3 cm AAA)
   4. If ≥3 cm aneurysm, record exact size and outcome in time (surveillance, treatment, no treatment)
   5. If treated, record treatment type (EVAR or Open) and outcome

ELIGIBILITY:
Inclusion Criteria:

* male and female patients
* peripheral arterial disease (ankle brachial index < 0,90 and/or reduction of > 0.15 after exercise test) or a carotid stenosis (stenosis ≥ 50%)
* age > 55 year

Exclusion Criteria:

* Patients unfit for endovascular or open surgery (as judged by vascular surgeon)
* Failure to master the dutch language

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral arterial disease or carotid arterial disease
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
AAA prevalence | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, Netherlands